CLINICAL TRIAL: NCT04226651
Title: Does Virtual Reality Exposure Therapy Affect Children's Dental Anxiety, Pain, and Behaviour? A Randomized, Placebo-Controlled Cross-Over Trial
Brief Title: The Effectiveness of Audiovisual Distraction Behavior Guidance Technique in Children With Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, BURAK BULDUR, Associate Prof., Cumhuriyet University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DIS-217
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Dental Anxiety; Dental Pain and Sensation Disorder
MeSH Terms: conditions — Toothache; Sensation Disorders | interventions — Eye Protective Devices

STUDY DESIGN:
Intervention Model Description: randomized, two-armed, within-subject, cross-over, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First dental visit (Active Comparator): Virtual Reality Exposure Therapy
  Interventions: Device: Virtual Reality Device
- Second Dental Visit (Placebo Comparator): Protective Glasses
  Interventions: Device: Protective glasses

INTERVENTIONS:
Device: Virtual Reality Device — The Virtual Reality system (PlayStation 4 VR, Sony Inc.) is a simple and easy to use distraction device. The system consists of a screen mounted on a binocular headset connected to a console or personal computer. The head-mounted display provides a high-resolution visual display and unmutes the sound from the headphones using a soundproof mechanism that provides clear sound.
  Arms: First dental visit
Device: Protective glasses — Each patient was informed about the dental procedure and was provided with protective glasses. All patients were told that they were wearing these glasses to ensure a pain- and stress-free treatment, and that the dentist would devote additional attention to the treatment.
  Arms: Second Dental Visit

SUMMARY:
This randomized, two-armed, placebo-controlled, cross-over, controlled trial aimed to evaluate the effect of virtual reality exposure therapy (VRET) on dental anxiety, pain, and behaviour among children undergoing dental treatment under local anaesthesia. The null hypotheses were as follows: VRET has no effect on reducing dental anxiety and dental pain scores of participants; and there is no difference between subjective and objective measure scores of dental anxiety and pain when VRET and attention palcebo-controlled (APC) groups are used to reduce anxiety in children undergoing dental treatment with local anaesthesia.

DETAILED DESCRIPTION:
This randomized, two-armed, placebo-controlled, cross-over, controlled trial adhered to the principles of the Declaration of Helsinki, good clinical practice guidelines, and applicable regulatory requirements. Ethics approval was obtained from the Health Ethics Committee of Sivas Cumhuriyet University (Sivas, Turkey; ID: 2018-02/08). All parents or guardians of children were educated about the study before enrollment and provided informed written consent to participate. The trial adhered to the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

The parameters used to calculate the sample size included a 95% confidence interval (CI), 80% statistical power, and a standard deviation of 1.90; accordingly, at least 64 subjects were required. This number was adjusted to 76 subjects to compensate for a projected loss of approximately 20% during follow-up. Thus, 76 healthy subjects between 7 and 11 years of age were included in the study. Participants who fulfilled the following criteria were included: systemically and mentally healthy; required restorative treatment for first mandibular permanent molar tooth with dentin caries in each mandibular quadrant with a bilateral inferior alveolar nerve block; absence of co-operative disability; and Frankl Scale score 2 or 3 during first dental examination. Patients with systemic or mental illnesses, reduced audiovisual capabilities, acute dental pain or trauma, those with previous painful or negative dental experience, and those who were extremely uncooperative were excluded.

The present randomized, two-armed, within-subject, cross-over, controlled trial included patients who applied to Department of Pediatric Dentistry, Cumhuriyet University, for routine dental treatment.The study comprised three visits: V0, baseline dental examination and inclusion; V1, first restorative treatment session; and V2, second restorative treatment session for symmetrical teeth. The initial oral and radiographic examination and Frankl Behaviour Scale scoring of all patients were performed by one experienced and pre-calibrated researcher. A dental assistant not participating in the study used a random-order generator (http://www.random.org) to randomize patients to the experimental group according to block randomization.

Eligible participants were treated in two different appointments: protective glasses only, without distraction (APC); or with the treatment condition (VRET). All procedures were performed by a single experienced and calibrated paediatric dentist (BB).

Participants were randomly assigned by a computer algorithm to receive VR with the first or second sequential dental treatment session and with protective glasses for the other treatment session. The investigators were blinded to treatment sequence until before the first dental treatment was to begin. Before VRET, the VR headset was shown to the patients, who were permitted to handle it. This enabled the patient to recognize the device and be familiar with it before treatment. Before starting treatment, the VR headset was placed on each patient's head, and the patient was asked whether the device caused pain or discomfort, and the patient's consent was confirmed. In the APC group, each patient was informed about the dental procedure and was provided with protective glasses. All patients were told that they were wearing these glasses to ensure a pain- and stress-free treatment, and that the dentist would devote additional attention to the treatment. This aimed to provide the patient with feeling like being in an experimental session. The reason for choosing an APC group with the routine protective glasses without distraction was to mitigate possible Hawthorne effects.

Regardless of experimental group, in the first treatment session, the mandibular first permanent molar tooth of each patient was restored with composite filling under local anaesthesia, while the opposite symmetrical tooth was treated in the second session. The duration of treatment in each session was noted and defined as the time from the subject sat on the chair to occlusal adjustment of restoration. First, the teeth were cleaned using fluoride-free prophylactic paste. The preparation was limited to removal of the caries, followed by rounding of the inner line and point angles. Cavity preparation was performed using an 80 µm grit diamond bur and completed using a 25 µm grit diamond bur (Intensiv, Viganello-Lugano, Switzerland). Isolation and contamination were controlled with suction and cotton rollers. In cases for which this was not sufficient, a rubber dam was used. Metal matrix bands and wooden wedges were also used where necessary.

Statistical analyses were performed using SPSS version 22.0 (IBM Corporation, Armonk, NY, USA). Descriptive analysis was used to summarize demographic characteristics and responses of the participants on each scale. The chi-squared test was used to compare age and sex differences at baseline. Repeated measures ANOVA was performed to analyse changes according treatment group, dental visit sequence and time point of treatment procedure. Differences with p < 0.05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Requiring restorative treatment for first mandibular permanent molar tooth with dentin caries in each mandibular quadrant with a bilateral inferior alveolar nerve block
* Co-operative ability

Exclusion Criteria:

* Systemic or mental illnesses
* Limited audiovisual capabilities
* Acute dental pain or trauma

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2019-09-16 (Actual)

PRIMARY OUTCOMES:
Dental Anxiety | Time 0: a minute after sitting in the dental unit ; Time 1: 1 min before local anaesthesia; Time 2: 1 min after local anaesthesia; Time 3: 1 min before end of the treatment
  Dental anxiety will be assessed using the Heart Rate with a portable pulse oximetry device
Dental Anxiety | Visit 0: 5 min before first inclusion visit, Visit 1: 5 min before first dental treatment visit,Visit 2: 5 min before second dental treatment visit,
  Dental anxiety was assessed using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) and Facial Image Scale (FIS)

SECONDARY OUTCOMES:
Dental Pain | Time 0: a minute after sitting in the dental unit ; Time 1: 1 min before local anaesthesia; Time 2: 1 min after local anaesthesia; Time 3: 1 min before end of the treatment
  Dental pain will be assessed using the Heart Rate with a portable pulse oximetry device
Dental Pain | Time 2: 1 min after local anaesthesia; Time 3: 1 min before end of the treatment
  Dental pain will be assessed using the Wong-Bakers Faces Pain Scale (WBS)
Dental behavior | Time 3: 1 min before end of the treatment
  Dental pain will be assessed using the Frankl Behaviour Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Burak Buldur, Sivas, Kampus, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not planned yet.